CLINICAL TRIAL: NCT01243710
Title: A Randomised Controlled Trial of Taurolidine With Heparin for Prevention of Recurrence of Catheter Related Bacteraemia in Haemodialysis Patients.
Brief Title: Taurolidine in Haemodialysis Catheter Related Bacteraemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUNN1007
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Renal Dialysis; Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taurolidine with heparin (Experimental)
  Interventions: Device: Taurolidine with heparin (500 units/ ml)
- Heparin (Active Comparator)
  Interventions: Device: Taurolidine with heparin (500 units/ ml)

INTERVENTIONS:
Device: Taurolidine with heparin (500 units/ ml) — Central venous catheter will be locked (the designated volume required to fill the dead space) with taurolidine with heparin after each dialysis session. The control arm will be locked with heparin as is current practice.
  Other Names: Taurolock Hep500

SUMMARY:
The purpose of this study is to determine whether taurolidine with heparin locking solution prevents recurrence of central venous catheter related blood stream infections in haemodialysis patients.

DETAILED DESCRIPTION:
Infections related to long-term haemodialysis catheters are associated with significant morbidity. A high proportion of those people initially treated with antibiotics to clear a catheter infection develop a second infection within six months, necessitating the removal and replacement of the dialysis catheter.

This study will examine the efficacy of an antimicrobial catheter locking solution called taurolidine with heparin in preventing a second infection within six months of a significant infection. This solution will be compared with the solution used currently (heparin) which is left inside the catheter between dialysis sessions.

This is a clinical study given that antimicrobial catheter locks are thought to reduce the risk of blood stream infections and the ultimate need for catheter change. However, there is concern that the absence of an anticoagulant in the lock solution increases the risk of catheter thrombosis, again requiring a change of catheter but for a separate reason. It is unclear therefore whether a solution containing both taurolidine (an antimicrobial) and heparin (an anticoagulant) will increase catheter survival.

The results of this study will help guide the appropriate suse of locking solutions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis patients established on dialysis for greater than 90 days who dialyse in-centre at any of the satellite dialysis units of Imperial College Healthcare NHS Trust
* All patients with a recent catheter related bacteraemia with an identified organism grown on microbiological culture and treated without catheter removal will be eligible for inclusion.

Exclusion Criteria:

* Those individuals in whom attempted catheter salvage is clinically not indicated.
* Unable to provide informed consent
* Known allergy to sodium citrate, heparin or taurolidine.
* Bleeding diathesis or physical cause for active bleeding.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Duration of bacteraemia-free catheter survival | Catheter survival measured up to six months from enrollment date.

SECONDARY OUTCOMES:
Catheter related flow problems | Catheter survival measured up to six months from enrollment date.
  Quantified by use of:
  1. Urokinase locks
  2. Systemic urokinase infusions
Hospital admissions for catheter related problems including catheter removal | Catheter survival measured up to six months from enrollment date.
Erythropoietin resistance | Catheter survival measured up to six months from enrollment date.
  Quantified by:
  1. Erythropoietin dose
  2. Number of blood transfusions required
Haemodialysis adequacy | Catheter survival measured up to six months from enrollment date.
  Quantified by:
  1. Kt/V
  2. Blood flows

CONTACTS AND LOCATIONS:
Overall Officials: Neill Duncan, MBBS, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom